CLINICAL TRIAL: NCT05142098
Title: Comparison of the Anti-Inflammatory Efficacy of Preemptive Dexamethasone and Etoricoxib Following Impacted Third Molar Surgery
Brief Title: Comparison of the Anti-Inflammatory Efficacy of Preemptive Dexamethasone and Etoricoxib
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hassan Hafeez, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hassan321
Record Dates: First submitted 2021-10-21; First posted 2021-12-02 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Dexamethasone; Glucocorticoids; Etoricoxib; Cyclooxygenase 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 4mg will be injected intramuscularly into the pterygomandibular space after achieving effective inferior dental block.
  Interventions: Drug: Dexamethasone
- Etoricoxib (Experimental): 2 tablets 60mg each would be given orally one hour prior to the surgery.
  Interventions: Drug: Etoricoxib 60 mg

INTERVENTIONS:
Drug: Dexamethasone — Intramuscular
  Other Names: Glucocorticoid
  Arms: Dexamethasone
Drug: Etoricoxib 60 mg — Orally
  Other Names: Cox-2 Inhibitor
  Arms: Etoricoxib

SUMMARY:
Impaction of mandibular third molars is a commonly encountered problem in oral surgery; patients frequently visit dental OPDs with complains related to the impacted molars, and in almost all situations, surgical removal of these impactions is the definitive treatment provided to such patients. This type of surgery often involves osteotomies and tooth sectioning, that initiates acute inflammatory responses which results in significant amount of postoperative discomfort owing to the associated pain, swelling and trismus; which considerably affects the quality of life that may span from days up to weeks in few instances. In the past decades, different group of medications have been used to counter these adverse postoperative sequelae, such as steroidal anti-inflammatory drugs (SAIDs) and non-steroidal anti-inflammatory drugs (NSAIDs).

MATERIAL AND METHODS:

Study design: Randomized, double-blind, clinical trial with a split-mouth design.

Setting: The study would be conducted at Oral & Maxillofacial Surgery department, Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences, Dow University of Health Sciences, Karachi.

Duration of study: Six months after the approval of synopsis. Sample size: A total of 170 patients would be included in the study, i.e. 85 in each group with 2 patients as a drop out.

Calculated sample size is 83 patients per group; utilizing Pass version 11 software with 95% confidence interval, mean ± S.D of swelling in dexamethasone group1 95.7 ± 11.1 and in etoricoxib group1 100.0 ± 8.3 at measurement 5.

Sampling technique: Purposive non-probability sampling technique would be used for the selection of patients.

Sample selection: Patients meeting the following criteria would be included in the study: 1. Age 18-35 years. 2. Absence of any systemic disease. 3. Mandibular third molars in similar position with similar root formation. 3. No use of any medication in last 03 days. 4. Absence of allergy to any drug used in the study. 5. Surgical site with no current signs or symptoms of infection.

Patients meeting any of the following criteria would be excluded from the study: 1. Pregnancy or lactation. 2. History of gastrointestinal bleeding or peptic ulcer. 3. Current smoking habit.

DETAILED DESCRIPTION:
Impaction of mandibular third molars is a commonly encountered problem in oral surgery; patients frequently visit dental OPDs with complains related to the impacted molars, and in almost all situations, surgical removal of these impactions is the definitive treatment provided to such patients. This type of surgery often involves osteotomies and tooth sectioning, that initiates acute inflammatory responses which results in significant amount of postoperative discomfort owing to the associated pain, swelling and trismus; which considerably affects the quality of life that may span from days up to weeks in few instances. In the past decades, different group of medications have been used to counter these adverse postoperative sequelae, such as steroidal anti-inflammatory drugs (SAIDs) and non-steroidal anti-inflammatory drugs (NSAIDs).

Owing to its predominant glucocorticosteroid effects, minimal sodium retention activity and long half-life, dexamethasone remains the most popular drug used in third molar surgery. And with the advantages of fewer gastrointestinal side effects, not disturbing platelet function and being well tolerated, the selective COX-2 inhibitor, Etoricoxib, is a suitable analgesic for the treatment of acute pain.

Lima et al2 concluded in their study that preemptive administration of dexamethasone showed better control of pain and swelling following impacted third molar extraction. Gaetano et al3 showed a greater reduction in incidence and severity of postoperative pain treated with etoricoxib compared with diclofenac, in impacted third molar surgery. Despite a lot of research related to the efficacy of dexamethasone and etoricoxib as preemptive drugs in controlling the postoperative sequelae, there is a negligible amount of research material available comparing the efficacy of these two anti-inflammatory drugs, therefore, the purpose of this study is to compare the preemptive anti-inflammatory effects of dexamethasone administered intramuscularly into the medial pterygoid muscle immediately after local anesthesia, with Etroicoxib given orally 1 hour prior to the surgery.

RATIONALE:

This study would help the clinicians in better understanding the anti-inflammatory consequences associated with a common oral surgical procedure. The results of this study would greatly enhance understanding about which drug to prescribe for the better control of anti-inflammatory sequelae of impacted third molar surgery, thereby, avoiding unnecessary drug prescriptions which would be ultimately beneficial for the patient undergoing treatment.

OBJECTIVE: The purpose of this study is to compare the preemptive anti-inflammatory efficacy of dexamethasone administered intramuscularly with etoricoxib given orally, following the impacted third molar surgery.

MATERIAL AND METHODS:

Study design: Randomized, double-blind, clinical trial with a split-mouth design.

Setting: The study would be conducted at Oral & Maxillofacial Surgery department, Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences, Dow University of Health Sciences, Karachi.

Duration of study: Six months after the approval of synopsis. Sample size: A total of 170 patients would be included in the study, i.e. 85 in each group with 2 patients as a drop out.

Calculated sample size is 83 patients per group; utilizing Pass version 11 software with 95% confidence interval, mean ± S.D of swelling in dexamethasone group1 95.7 ± 11.1 and in etoricoxib group1 100.0 ± 8.3 at measurement 5.

Sampling technique: Purposive non-probability sampling technique would be used for the selection of patients.

Sample selection: Patients meeting the following criteria would be included in the study: 1. Age 18-35 years. 2. Absence of any systemic disease. 3. Mandibular third molars in similar position with similar root formation. 3. No use of any medication in last 03 days. 4. Absence of allergy to any drug used in the study. 5. Surgical site with no current signs or symptoms of infection.

Patients meeting any of the following criteria would be excluded from the study: 1. Pregnancy or lactation. 2. History of gastrointestinal bleeding or peptic ulcer. 3. Current smoking habit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35 years.
2. Absence of any systemic disease.
3. Mandibular third molars in similar position with similar root formation.

3. No use of any medication in last 03 days. 4. Absence of allergy to any drug used in the study. 5. Surgical site with no current signs or symptoms of infection.

Exclusion Criteria:

1. Pregnancy or lactation.
2. History of gastrointestinal bleeding or peptic ulcer.
3. Current smoking habit.
4. Patient encountering any complication during/after procedure.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
assessment of post operative complications after dexamethasone | within one week after procedure
  dexamethasone is more effective in controlling post operative pain, swelling and trismus following impacted third molar surgery.
assessment of post operative complications after etoricoxib | within one week after procedure
  Etoricoxib is more effective in controlling post operative pain, swelling and trismus following impacted third molar surgery.

CONTACTS AND LOCATIONS:
Overall Officials: hassan hafeez, Principal Investigator — DUHS

IPD SHARING:
Plan to Share IPD: No